CLINICAL TRIAL: NCT06858033
Title: Assessment of the Effect of Labio-Lingual Spring Hawley and Clear Aligners on Children's Oral Microflora and Salivary Parameters
Brief Title: Evaluation of the Effect of Labio-Lingual Spring Hawley and Clear Aligners on Periodontal Health and Salivary Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozge Gungor (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Sponsor-Investigator, Ozge Gungor, pHd, DDS, Assoc. Prof. Dr. Pediatric Dentist, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AkdenizUıremkapıcı001
Record Dates: First submitted 2025-01-20; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Anterior Crossbite
Keywords: Clear aligner; Labiolingual spring hawley; Oral health
MeSH Terms: interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clear aligner users (Experimental): Patients who were treated with clear aligners were referred to as 'clear aligner users'.
  Interventions: Device: Clear aligner
- Labiolingual spring hawley users (Experimental): Patients who were treated with clear aligners were referred to as 'Labiolingual spring hawle users'.
  Interventions: Device: Labiolingual spring hawley

INTERVENTIONS:
Device: Clear aligner — The effects of treatment on periodontal parameters (plaque index, gingival index, bleeding index on probing), salivary parameters (stimulated/unstimulated flow rate, stimulated/unstimulated pH, buffering capacity) and oral microorganism counts (S. mitis, S. salivarius, S. mutans, C. albicans) of children treated with labiolingual spring hawley and clear aligners were investigated.
  Arms: Clear aligner users
Device: Labiolingual spring hawley — The effects of treatment on periodontal parameters (plaque index, gingival index, bleeding index on probing), salivary parameters (stimulated/unstimulated flow rate, stimulated/unstimulated pH, buffering capacity) and oral microorganism counts (S. mitis, S. salivarius, S. mutans, C. albicans) of children treated with labiolingual spring hawley and clear aligners were investigated.
  Arms: Labiolingual spring hawley users

SUMMARY:
Objective: The aim of our study was to determine the effect of two different types of removable appliances on periodontal health, dental plaque colonization, as well as saliva, pH, flow rate, and buffering capacity of the patients.

Method: A total of 30 pediatric patients aged 7-12 years were treated with a total of 30 appliances including 15 clear aligners (Group A) and 15 labiolingual spring hawleys (Group B). In the clinical examination of the patients, dental caries status was evaluated by DMFT and dft index, periodontal health status was evaluated by probing pocket depth measurements and plaque, gingival and probing bleeding indices. In addition, saliva and dental plaque samples were taken and salivary parameters and microbiologic structure of plaque were analyzed. All these procedures were performed in 2 different time periods for each patient; before and after the treatment. The results were statistically evaluated using SPSS (SPSS Statistics v23.0 for Windows, Chicago, IL, USA).

DETAILED DESCRIPTION:
In the clinical examination of the participants, dental caries status was evaluated by DMFT and dft index, and periodontal health status was evaluated by probing pocket depth measurements; PI, GI, SDI. In addition, saliva and dental plaque samples were taken and salivary parameters (flow rate, pH and buffering capacity) and microbiological structure of plaque were analyzed.

ELIGIBILITY:
Inclusion Criteria:

• Dental anterior crossbite

Exclusion Criteria:

* Skeletal anterior crossbite
* Systemic disease
* Regular medication use

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
PIaque index (PI) | 3 months
  Based on Silness-Löe (1963, 1967) PI values, bacterial plaque and plaque thickness in direct contact with the marginal gingiva are evaluated. The evaluation is made with the Williams-marked University of Michigan 'O' periodontal probe, and PI values are recorded from a total of 4 surfaces of each tooth included in the study, namely mesial, distal, buccal and lingual. The averages of these values are calculated for each patient. The average scores obtained are evaluated in the 0-3 score range. An increase in the calculated scores indicates that periodontal health is negatively affected.
DMFT index | 3 months
  To determine the DMFT index score, decayed teeth in permanent teeth are indicated as "D", lost teeth extracted due to decay are indicated as "M", and filled teeth are indicated as "F". The DMFT index is calculated by adding the D, M, F values and dividing them by the total number of permanent teeth. An increase in the calculated scores indicates that oral and dental health is negatively affected.
Oral microorganisms count | 3 months
  S. mitis, S. salivarius, S.mutans, C. albicans (cfu/ml)
Gingival index (GI) | 3 months
  The degree of gingivitis is assessed using the Silness-Löe (1963, 1967) GI. The average of the measurements taken from four sides of the tooth determines the GI score of the tooth, and the average of the measurements of all teeth determines the individual's gingival index score. The scores obtained are evaluated in the range of 0-3. An increase in the calculated scores indicates that periodontal health is negatively affected.
Bleeding on probing index (BOP) | 3 months
  In order to determine the inflammatory status of the pocket base and pocket epithelium, a score is given as positive (+) or negative (-) according to whether there is bleeding in the sulcus 20 seconds after the pocket depth measurement from a total of 4 surfaces of the teeth, mesial, distal, buccal and lingual. BOP is calculated as a score by dividing the number of bleeding teeth by the total number of tooth surfaces in each patient. An increase in the calculated scores indicates that periodontal health is negatively affected.
dft index | 3 months
  The dft Index is the calculated form of the DMFT index for primary teeth. When calculating the dft group index, missing teeth are not included in the calculation. Because it is difficult to diagnose the reason for the loss of primary teeth and there is a high probability of error. For this reason, the number of decayed and filled teeth is calculated during the examination. Decayed teeth are indicated with "d" and filled teeth with "f". The dft index is calculated by adding the d and f values and dividing them by the total number of permanent teeth. An increase in the calculated scores indicates that oral and dental health is negatively affected.

CONTACTS AND LOCATIONS:
Overall Officials: Özge GÜNGÖR, DDS, Assoc. Prof. Dr., Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University Faculty of Dentistry, Department of Pediatric Dentistry, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapicii I, Erken Gungor O, Yildirim K, Atas C, Yilmaz Coban A. Impact of Z-spring appliance and clear aligner therapy on oral microorganisms in children: A clinical trial. Saudi Med J. 2025 Jul;46(7):825-830. doi: 10.15537/smj.2025.46.7.20250264. PMID 40628430